CLINICAL TRIAL: NCT04035707
Title: Serum Tryptase Concentration During General Anaesthesia With Rocuronium
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Bialystok (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 143-14548/14
Record Dates: First submitted 2019-07-11; First posted 2019-07-29 (Actual); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Hypersensitivity Reaction
Keywords: general anaesthesia; mast cell; rocuronium; tryptase
MeSH Terms: conditions — Hypersensitivity | interventions — Rocuronium

STUDY DESIGN:
Intervention Model Description: The study included 126 women given a general volatile anesthesia: group I - 66 - using the rocuronium and group II - 60 - without neuromuscular relaxants. Informations about perioperative fluid therapy and doses of rocuronium were noticed. The blood samples were collected to perform tryptase concentration analysis: preoperatively - before anesthesia and postoperatively - after recovery from anesthesia.
Who Masked: Investigator
Masking Description: qualification according surgical operation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- anaesthesia with rocuronium (Experimental): rocuronium is used during anaesthesia
  Interventions: Drug: Rocuronium; Drug: general volatile anaesthesia
- anaesthesia without rocuronium (Experimental): during anaesthesia rocuronium is not used
  Interventions: Drug: general volatile anaesthesia

INTERVENTIONS:
Drug: Rocuronium — using rocuronium as a relaxants during general anaesthesia
  Arms: anaesthesia with rocuronium
Drug: general volatile anaesthesia — method of anaesthesia

SUMMARY:
Rocuronium is a aminosteroid structured, non-depolarizing neuromuscular blocking agents (NMB). Epidemiological data presents that the frequency of hypersensitivity reactions caused by rocuronium have been increased. Determinations of serum tryptase concentrations are interdisciplinary recommended in diagnosis of its adverse reactions. No studies have been performed to explain specific role of rocuronium doses on serum tryptase values. The aim of this study was to investigate the potential effect of rocuronium on serum tryptase concentrations.

DETAILED DESCRIPTION:
The greatest risk of hypersensitivity occurs during anesthesia for female patients and it is connected with the induction phase using skeletal muscle relaxants . Epidemiological data presents that the frequency of hypersensitivity reactions caused by rocuronium have been increased. Due to the multiple advantages reports of triggering allergic or hypersensitivity reactions caused by rocuronium create doubts about the safety of application .

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-2, no allergy and perioperative hypersensitivity reactions during anaesthesia

Exclusion Criteria:

* steroid therapy, allergy in medical history, mastocytosis

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2009-06-25 (Actual); Primary Completion 2010-06-25 (Actual); Study Completion 2014-05-15 (Actual)

PRIMARY OUTCOMES:
tryptase | up to 40 minutes after surgery
  serum tryptase concentration

CONTACTS AND LOCATIONS:
Overall Officials: Urszula Kosciuczuk, Principal Investigator — Medical University in Bialystok

IPD SHARING:
Plan to Share IPD: No
IPD are available only for investigators

REFERENCES:
- [Derived] Kosciuczuk U, Knapp P, Jakubow P. Effect of body mass index and rocuronium on serum tryptase concentration during volatile general anesthesia: an observational study. Clinics (Sao Paulo). 2020;75:e1701. doi: 10.6061/clinics/2020/e1701. Epub 2020 Aug 10. PMID 32785569